CLINICAL TRIAL: NCT07086898
Title: Impact of Adding Integrated Neuromuscular Inhibition Technique to Postural Correction Exercises in Patients With Cervicogenic Headache
Acronym: CGH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, principle investigator : alshaymaa shaaban abd el azeim, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005850
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Cervicogenic Headache
Keywords: integrated neuromuscular inhibition technique; postural correction exercises; cervicogenic headache
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Intervention Model Description: integrated neuromuscular inhibition technique and postural correction exercises
Who Masked: Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Neuromuscular Inhibition Technique (Experimental): Forty-five patients will receive integrated neuromuscular inhibition technique plus postural correction exercises three times a week for six weeks
  Interventions: Other: Integrated Neuromuscular Inhibition Technique; Other: Postural Correction Exercise
- Postural Correction Exercise (Active Comparator): Forty-five patients will receive postural correction exercises three times a week for six weeks
  Interventions: Other: Postural Correction Exercise

INTERVENTIONS:
Other: Integrated Neuromuscular Inhibition Technique — Patients will receive integrated neuromuscular inhibition technique in the form of intermittent ischemic compression, strain counterstrain, and muscle energy technique plus postural correction exercises
  Arms: Integrated Neuromuscular Inhibition Technique
Other: Postural Correction Exercise — The exercise program will be in the form of stretching exercises for the sternocleidomastoids (SCM), the scalenes, and upper fibers of trapezius; strengthening isometric exercises for the neck flexors, extensors, lateral flexors, and neck rotators; and postural correction exercises.

SUMMARY:
this study will be conducted to investigate the impact of adding integrated neuromuscular inhibition technique to postural correction exercises in patients with cervicogenic headache

DETAILED DESCRIPTION:
Cervicogenic headache (CeH) is a secondary headache attributed to dysfunctions of the cervical spine. CGH is a non-throbbing, unilateral, side locked headache that originates in the cervical spine and gradually spreads to the occipital, temporal and orbital areas. It is associated with neck pain or stiffness and is often aggravated by sustained neck postures, repeated neck movements or physical activity. INIT is effective as it causes sustained or intermittent compression which causes ischemia reduces local circulation until pressure is released, after which a flushing of fresh oxygenated blood occurs. Mechanoreceptors impulses interface with slower pain messages reducing amount of pain messges reaching the brain, releasing pain relieving hormones, decreasing myofascial pain. Stretches the taut bands of muscles fibers. INIT along with strengthening excercises proved to be beneficial in decreasing disability improving Range of motion.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 60 years old patient with unilaterally of the head pain
* pain triggered by external pressure over the upper cervical joints (c1-c3)
* pain elicited by the neck movements, and/or sustained awkward positions with reduced neck ROM
* headache intensity pain score of at least 20mm on the Visual analogue scale (VAS)
* headache frequency of at least once a week for at least 3 months
* minimum neck disability index score of 10 points or greater

Exclusion Criteria:

* Migraine, tension- type headache, tumor, osteoporosis, fracture, rheumatoid arthritis and metabolic diseases.
* Prolonged history of steroid use.
* Resting blood pressure greater than 140/90 mmhg.
* cervical spinal stenosis, diminished sensation and central nervous system involvement,
* previous

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
pain intensity | up to six weeks
  visual analogue scale will be used to asses pain intensity which patient will be instructed to put point on line from no pain to tolerable pain. The scale consists of a line, usually 100 mm long, ranging from no pain or discomfort (zero) , to the worst pain that could possibly feel .
headache disability | up to 6 weeks
  The Headache spesific Disability Questionnaire was used to assess headcahe disability. it is a self-administered scale with 9 items that assesses pain intensity, work or school disruptions, and the effect on recreational activities in individuals with headache complaints. Higher scores reflect greater impairment.

SECONDARY OUTCOMES:
pressure pain threshold | up to 6 weeks
  pressure pain threshold pressure pain threshold will be assessed by commander algometer
cervical range of motion | up to 6 weeks
  range of motion will be measured by inclinometer CROM. The CROM (deluxe version - Performance Attainment Associates, Roseville, MN, USA) measures the cervical range of motion5- for fexion, extension, lateral fexion, and rotation using separate inclinometers. These inclinometers are attached to a frame similar to that for eyeglasses one in the sagittal plane for fexion - extension, second in the frontal plane for lateral fexion and a third in the horizontal plane for rotation.
headache frequency | up to six weeks
  the number of days the subjects feel headache (headache frequency).
medication intake | up to six weeks
  from the patients' diary in the last week , medications intake will be recorded as follow: 1) not at all; 2) once a week; 3) once every couple of days; 4) once or twice a day; or 5) three or more times a day
headache duration | up to six weeks
  the total hours of headache (headache duration).